CLINICAL TRIAL: NCT03063112
Title: Comparative Study Between Radiofrequency Thermocoagulation and Chemical Neurolysis of Thoracic Splanchnic Nerve Bilaterally for the Management of Abdominal Cancer Pain
Brief Title: Radiofrequency and Chemical Neurolysis of Thoracic Splanchnic Nerve for Abdominal Cancer Pain
Acronym: RF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Fatma Al Zahraa Hamed Abdel Hameed, Lecturer of anasthesia and pain relief, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Ethical committee 167
Record Dates: First submitted 2017-02-10; First posted 2017-02-24 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Abdominal Cancer
MeSH Terms: interventions — Lidocaine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1( radiofrequency group ) (Active Comparator): Bilateral thoracic splanchnic nerves block will be performed by radiofrequency thermocoagulation at two level of vertebra T10 and T11 by using radiofrequency generator device and lidocaine 2% before thermal lesion
  Interventions: Device: Radiofrequency generator device; Drug: Lidocaine
- Group 2 ( alcohol group ) (Placebo Comparator): Bilateral thoracic splanchnic nerves block will be performed by ethyl alcohol at one level of vertebraT11 by using of C arm fluoroscopic device.
  Interventions: Device: C arm fluoroscopic device; Drug: Ethyl alcohol

INTERVENTIONS:
Device: Radiofrequency generator device — sympathetic blockade or ablation of thoracic splanchnic nerves
  Other Names: Physical neurolysis
  Arms: Group 1( radiofrequency group )
Drug: Lidocaine — sympathetic blockade or ablation of thoracic splanchnic nerves
  Arms: Group 1( radiofrequency group )
Device: C arm fluoroscopic device — sympathetic blockade or ablation of thoracic splanchnic nerves
  Arms: Group 2 ( alcohol group )
Drug: Ethyl alcohol — sympathetic blockade or ablation of thoracic splanchnic nerves
  Other Names: Chemical neuolysis
  Arms: Group 2 ( alcohol group )

SUMMARY:
The study compares between the efficacy, safety and impact on the quality of life of radiofrequency thermocoagulation and chemical neurolysis of bilateral thoracic splanchnic nerves in the management of refractory pain which developed in patients suffering from upper abdominal cancer.

DETAILED DESCRIPTION:
Radiofrequency thermocoagulation of splanchnic nerves was done bilaterally at level of thoracic vertebra T10 and T11 ( there were no enough studies done to test the efficacy, safety and impact on the quality of life of radiofrequency thermocoagulation of splanchnic nerves at level of T10 ). Aim of the Study is to compare between the efficacy, safety and impact on the quality of life of radiofrequency thermocoagulation of bilateral thoracic splanchnic nerves at level T10 and T11 vertebra and chemical neurolytic block of them at level of T11 vertebra only in the management of upper abdominal cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from upper abdominal cancer pain.
2. Visceral pain with visual analogue pain score ≥ 4.
3. Normal coagulation profile.
4. Positive diagnostic test.
5. Written informed consent from the patients .

Exclusion Criteria:

1. Patients with organ failure.
2. Coagulation disorders.
3. Local infection at the puncture site or sepsis.
4. Allergy to the contrast dye or alcohol.
5. Severe displacement of intra-abdominal structures.
6. Pregnant women.
7. Documented metastatic lesions.
8. Psychiatric illness affecting cooperation.
9. De-compensated cardiac disorders.
10. Liver and renal dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-04-10 (Estimated); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 3 months
  Visual analogue pain scale

SECONDARY OUTCOMES:
Decrease the need for analgesic drugs | 3 months
  Reduction of total oral morphine consumption dose in mg per day

CONTACTS AND LOCATIONS:
Overall Officials: Samy A Erfan, Professor, Study Director — Head of the department
Locations (1):
- South Egypt Cancer Institute, Asyut, Assuit Governrate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided